CLINICAL TRIAL: NCT02980094
Title: Effects of Inclusion of Sunflower Oil, Vitamin E and Selenium in the Diet of Dairy Cows on Milk Composition and Its Influence on Nutrition and Health of Elderly
Brief Title: Milk Biofortification Promotes Health Benefits in Institutionalized Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eduardo Ferriolli (Other)
Responsible Party: Sponsor-Investigator, Eduardo Ferriolli, Assistant professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 4921/2011
Record Dates: First submitted 2016-11-09; First posted 2016-12-02 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Nutrient Deficiency; Age-Related Immunodeficiency; Vitamin E Deficiency; Selenium Deficiency; Fatty Acid Deficiency; Institutionalization; Disinhibited Attachment
Keywords: aging; nutrients; milk; dietary supplementation
MeSH Terms: conditions — Vitamin E Deficiency | interventions — Oils; Vitamin E; Selenium; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Milk Control group(C) (Placebo Comparator): Using a randomized block design, 25 institutionalized elderly to receive the milk 3 times per day produced by lactating cows fed with the following diet, one of the group is control (C), without vitamin E, selenium, sunflower oil in the cow's food.
  Interventions: Dietary Supplement: Milk Control group(C)
- Milk Antioxidant group(A) (Experimental): Using a randomized block design, 25 institutionalized elderly to receive the milk produced by lactating cows fed with the following diet: control (C) +vitamin E+ selenium (A).
  Interventions: Dietary Supplement: Milk Antioxidant group(A)
- Milk Oil group(O) (Experimental): Using a randomized block design, 25 institutionalized elderly to receive the milk produced by lactating cows fed with the following diets: control (C)+sunflower oil (O).
  Interventions: Dietary Supplement: Milk Oil group(O)
- Milk Antioxidant and oil(AO) (Experimental): Using a randomized block design, 25 institutionalized elderly to receive the milk produced by lactating cows fed with the following diets: control C+sunflower oil+vitamin E+selenium (AO) .
  Interventions: Dietary Supplement: Milk Antioxidant and oil(AO)

INTERVENTIONS:
Dietary Supplement: Milk Antioxidant group(A) — There is no intervention pre-specified before the institutionalized elderly to receive three times per day of milk (total 600ml of milk all day) produced by lactating cows fed with the following diets: control (C)+selenium and vitamin E (A).
  Other Names: add control diet(C) in the cow's food; add selenium in the cow's food; add vitamin E in the cow's food
  Arms: Milk Antioxidant group(A)
Dietary Supplement: Milk Oil group(O) — There is no intervention pre-specified before the institutionalized elderly to receive three times per day of milk (total 600ml of milk all day) produced by lactating cows fed with the following diets: control (C)+sunflower oil (O).
  Other Names: add control diet(C) in the cow's food; add sunflower oil group in the cow's food
  Arms: Milk Oil group(O)
Dietary Supplement: Milk Antioxidant and oil(AO) — There is no intervention pre-specified before the institutionalized elderly to receive three times per day of milk (total 600ml of milk all day) produced by lactating cows fed with the following diets:control (C)+selenium, vitamin E and sunflower oil (AO).
  Other Names: add control diet(C) in the cow's food; add selenium in the cow's food; add vitamin E in the cow's food; add sunflower oil in the cow's food
  Arms: Milk Antioxidant and oil(AO)
Dietary Supplement: Milk Control group(C) — There is no intervention pre-specified before the institutionalized elderly to receive three times per day of milk (total 600ml of milk all day) produced by lactating cows fed with the following diets: control (C)
  Other Names: add control diet (C) in the cow's food; without vitamin E in the cow's food; without selenium in the cow's food; without sunflower oil in the cow's food
  Arms: Milk Control group(C)

SUMMARY:
The project aims to study the effects of inclusion of sunflower oil, vitamin E and selenium in the diet of dairy cows on milk composition and the influence of modified milk on nutrition and health of elderly. To achieve those goals, two experiments will be conducted, both lasting 12 weeks. In the first one, 32 cows at the beginning of lactation will be allotted in a completely randomized block design with a 2 x 2 factorial arrangement of treatments, as follow: 1) control diet; 2) control diet plus selenium and vitamin E; 3) control diet plus sunflower oil diet; 4) control diet plus sunflower oil, selenium and vitamin E. This experiment seeks the development of modified milks through nutritional manipulation of cow's diet. Concomitantly, in the second experiment, 132 elderly people will receive the four different kinds of milk produced in the first experiment in a completely randomized block (gender) design. The selection of the elderly for each group shall be composed clinical evaluations. Will be conducted biochemical tests before and after supplementation of milk consumption (serum α-tocopherol, selenium, analysis of fatty acid profile). Assessment of nutritional status will be made body mass index (BMI) with each participant before and after the experiment of 12 weeks, including body composition by multifrequency bioelectrical impedance analysis (BIA), evaluating the strength of pressure of the hand portable dynamometer, demographics and food consumption. The study of human nutrition and health will be held in the form of a double-blind study. The second experiment aims to study nutrition and health of elderly people, as it is expected that milk produced with better fatty acid profile, vitamin and minerals can improve the inflammatory profile of markers of the elderly. This project is important for the human population in general, particularly elderly people, health workers, human and animal nutritionists, and especially for the milk chain, as it has a potential to develop new dairy products and boost milk consumption.

ELIGIBILITY:
Inclusion Criteria:

* Any institution residents that use milk in their usual diet.

Exclusion Criteria:

* Inability to drink
* Use of enteral diets
* Lactose intolerance
* Autoimmune disorders
* Infections, allergies or inflammation in the two weeks prior to blood collection.

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in serum α-tocopherol | before and after 12 weeks
  Assessment by blood sampling. Collect of α-tocopherol before and after to 12 weeks of milk supplementation
Change in serum selenium | before and after 12 weeks
  Assessment by blood sampling. Collect of selenium before and after to 12 weeks milk supplementation
Change in analysis of fatty acid profile | before and after 12 weeks
  Assessment by blood sampling. Collect of analysis of fatty acid profile before and after to 12 weeks of milk supplementation

SECONDARY OUTCOMES:
Assessment of nutritional status: food intake questionnaire | before and after 12 weeks
  Food consumption questionnaire during the milk supplementation
Change in handgrip strength | before and after 12 weeks
  Measure of the hand grip strength using a portable dynamometer before and after 12 weeks of milk supplementation
Assessment of nutritional status: anthropometry (BMI) | before and after 12 weeks
  BMI before and after 12 weeks of milk supplementation
Assessment of nutritional status: body composition | before and after 12 weeks
  Body composition measured by multifrequency bioelectrical impedance analysis (BIA) before and after to 12 week of milk supplementation
Assessment demographics: questionnaire | before and after 12 weeks
  Demographics questionnaire applied during the milk supplementation

OTHER OUTCOMES:
Change in profile of Inflammatory markers | before and after 12 weeks
  Serum Cytokines measured in blood sample before and after to 12 weeks of milk supplementation
Change in gene expression | before and after 12 weeks
  Gene expression of cyclooxygenase -1 (COX-1) e-2, monocyte chemotactic protein (MCP-1), peroxisome proliferator-activated receptor (PPAR) (-δ, -α and -β / δ) measured in blood sample before and after to 12 weeks milk supplementation
Change in production of reactive oxygen species | before and after 12 weeks
  Production of reactive oxygen species (ROS) produced by stimulated neutrophils measured in blood sample before and after to 12 weeks milk supplementation
Change in phagocytic activity | before and after 12 weeks
  Phagocytic activity measured in blood sample before and after to 12 weeks milk supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Ferriolli, PhD, Principal Investigator — Study Principal Investigator; Helio Vannucchi, PhD, Study Chair — Study Chair investigator
Locations (1):
- Clinics Hospital of the Ribeirao Preto Medical School, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barr SI, McCarron DA, Heaney RP, Dawson-Hughes B, Berga SL, Stern JS, Oparil S. Effects of increased consumption of fluid milk on energy and nutrient intake, body weight, and cardiovascular risk factors in healthy older adults. J Am Diet Assoc. 2000 Jul;100(7):810-7. doi: 10.1016/S0002-8223(00)00236-4. PMID 10916520
- [Result] Bouis HE, Hotz C, McClafferty B, Meenakshi JV, Pfeiffer WH. Biofortification: a new tool to reduce micronutrient malnutrition. Food Nutr Bull. 2011 Mar;32(1 Suppl):S31-40. doi: 10.1177/15648265110321S105. PMID 21717916
- [Result] Witkowska Z, Michalak I, Korczynski M, Szoltysik M, Swiniarska M, Dobrzanski Z, Tuhy L, Samoraj M, Chojnacka K. Biofortification of milk and cheese with microelements by dietary feed bio-preparations. J Food Sci Technol. 2015 Oct;52(10):6484-92. doi: 10.1007/s13197-014-1696-9. Epub 2015 Jan 21. PMID 26396393
- [Result] Kratz M, Baars T, Guyenet S. The relationship between high-fat dairy consumption and obesity, cardiovascular, and metabolic disease. Eur J Nutr. 2013 Feb;52(1):1-24. doi: 10.1007/s00394-012-0418-1. Epub 2012 Jul 19. PMID 22810464
- [Derived] Pfrimer K, Ferriolli E, Takeuchi PL, Salles MS, Saran-Netto A, Zanetti MA, Roma-Junior LC, Braga CBM, Domenici FA, Valim YM, Paschoalato AB, Marchi LF, Azzolini AE, Donadi EA, Martinez E, Vannucchi H. Effects of the Consumption of Milk Biofortified with Selenium, Vitamin E, and Different Fatty Acid Profile on Immune Response in the Elderly. Mol Nutr Food Res. 2018 Feb;62(4). doi: 10.1002/mnfr.201700307. Epub 2018 Jan 15. PMID 29193757